CLINICAL TRIAL: NCT05356156
Title: A Multicenter, Randomized, Controlled Clinical Trial of the Safety of Mesenteric Defects Closure After Radical Gastrectomy
Brief Title: The Safe Study of Routine Closure of Mesenteric Defects Versus Non-closure After Radical Gastrectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JSGCU-2203
Record Dates: First submitted 2022-04-23; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closure of the mesenteric defects (Experimental): Closure of the mesenteric defects will be performed after radical gastrectomy in patients with gastric or esophagogastric junction adenocarcinoma.
  Interventions: Procedure: Closure of the mesenteric defects
- Non-closure of the mesenteric defects (Active Comparator): Non-closure of the mesenteric defects will be performed after radical gastrectomy in patients with gastric or esophagogastric junction adenocarcinoma.
  Interventions: Procedure: Non-closure of the mesenteric defects

INTERVENTIONS:
Procedure: Closure of the mesenteric defects — The surgically created mesenteric defects will be closed after radical gastrectomy with D1+/D2 lymph node dissection.
  Arms: Closure of the mesenteric defects
Procedure: Non-closure of the mesenteric defects — The surgically created mesenteric defects will not be closed after radical gastrectomy with D1+/D2 lymph node dissection.
  Arms: Non-closure of the mesenteric defects

SUMMARY:
To compare the incidence of internal hernia, overall survival and short-term surgical safety of routine closure of the surgically created mesenteric defects versus non-closure for patients with adenocarcinoma of the gastric or esophagogastric junction who underwent radical gastrectomy (D1+/D2 lymph node dissection).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years；
* Primary lesion is diagnosed with endometrial biopsy as adenocarcinoma of the stomach or esophagogastric junction, including: papillary adenocarcinoma, tubular adenocarcinoma, mucinous adenocarcinoma, poorly cohesive carcinoma (including signet ring cell carcinoma and other variants), mixed adenocarcinoma, etc.；
* The gastric primary lesion is located in the antrum, body or fundus of stomach or the esophagogastric junction. It is expected that radical gastrectomy with D1+/D2 lymph node dissection achieves R0 resection (multiple primary cancers are also applicable)；
* BMI(Body Mass Index) < 30 kg/m2；
* No history of upper abdominal surgery (except for laparoscopic cholecystectomy)；
* No prior treatment of chemotherapy, radiotherapy, targeted therapy, immunotherapy, etc.；
* Preoperative ECOG (Eastern Cooperative Oncology Group) performance status score 0 or 1；
* Preoperative ASA (American Society of Anesthesiologists) scoring I-III；
* Sufficient vital organ functions；
* Signed informed consent.

Exclusion Criteria:

* Women during pregnancy or lactation；
* Suffer from other malignant tumors within 5 years；
* Preoperative body temperature ≥ 38°C or complicated with infectious diseases requiring systemic treatment；
* Severe mental illness；
* Severe respiratory disease；
* Severe liver and kidney dysfunction；
* History of unstable angina or myocardial infarction within 6 months；
* History of cerebral infarction or cerebral hemorrhage within 6 months；
* Continuous application of glucocorticoid within 1 month (except for topical application)；
* Accompanied by gastric cancer complications (bleeding, perforation, obstruction, etc.) ；
* The patient has participated in or is participating in other clinical studies (within 6 months).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1968 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
The incidence of internal hernia within 3 years after surgery | 3 years
  Internal hernia were identified by surgical exploration or abdominal computed tomography (CT) from surgical and medical records during the postoperative 3 years of follow-up.

SECONDARY OUTCOMES:
The incidence of intraoperative complications | up to 2 hours after surgery
  The intraoperative complications occur from the beginning of skin cutting to the completion of sewn skin, including surgical complications, anesthesia related complications and pneumoperitoneum related complications.
Incidence of postoperative intestinal obstruction | 3 years
  Refers to the incidence of postoperative intestinal obstruction observed during follow-up period.
Overall survival at 3 years after surgery | 3 years
  The overall survival of patients with gastric or esophagogastric junction adenocarcinoma are evaluated at 3 years after radical gastrectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Zekuan Xu, M.D., Ph.D., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China